CLINICAL TRIAL: NCT01707329
Title: A Phase II Randomised, Double Blind, Placebo Controlled Study to Assess the Efficacy and Safety of Icotinib in Combination With Chemotherapy Versus Chemotherapy Alone in Patients Who Have Progressed After Icotinib Treatment in NSCLC
Brief Title: Icotinib in Combination With Chemotherapy Versus Chemotherapy Alone in Patients Progressed After Icotinib Treatment
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Betta Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BD-IC-IV44
Record Dates: First submitted 2012-10-11; First posted 2012-10-16 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy; Docetaxel; Pemetrexed; icotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chemotherapy (Active Comparator): Docetaxel 60-75mg/m2, 4 cycles; or pemetrexed 500mg/m2, 4 cycles.
  Interventions: Drug: Chemotherapy
- Icotinib+Chemotherapy (Experimental): Icotinib: 125 mg is administered orally three times per day. Chemotherapy: docetaxel 75mg/m2, 4 cycles; or pemetrexed 500mg/m2, 4 cycles.
  Interventions: Drug: Icotinib+chemotherapy

INTERVENTIONS:
Drug: Chemotherapy — Docetaxel 60-75mg/m2, 4 cycles; or pemetrexed 500mg/m2, 4 cycles.
  Other Names: Taxotere; ALIMTA
  Arms: Chemotherapy
Drug: Icotinib+chemotherapy — Icotinib: 125 mg is administered orally three times per day. Chemotherapy: docetaxel 75mg/m2, 4 cycles; or pemetrexed 500mg/m2, 4 cycles.
  Other Names: Icotinib; Comana; BPI-2009
  Arms: Icotinib+Chemotherapy

SUMMARY:
This phase II randomised, double blind, placebo controlled, multicentre trial is designed to assess the efficacy and safety of continuous icotinib plus chemotherapy versus chemotherapy alone in patients who have progressed after benefiting from previous second or third-line icotinib treatment (more than 6 months) in locally advanced or metastatic non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed stage IIIB/IV lung cancer(exclude patients confirmed by sputum cytology)
* No previous targeted treatment such as gefitinib, erlotinib.
* With a measurable disease(longest diameters >=10mm with Spiral computed tomography (CT)and >=20mm with conventional CT) according to RECIST Criteria
* WHO performance status(PS)<= 2
* N>=1.5×109/L, Plt>=1.0×109/L,Hb>=10g/dL;AST&ALT should <3ULN(without liver metastasis) or <5ULN(with liver metastasis).TBIL<=1.5ULN.
* Signed and dated informed consent before the start of specific protocol procedures.

Exclusion Criteria:

* Allergic to icotinib
* Patients with metastatic brain tumors with symptoms.
* Experience of Anti-EGFR(the epidermal growth factor receptor) Monoclonal Antibody or small molecular compounds therapy such as gefitinib, erlotinib or Cetuximab.
* Severe systemic disease out of control such as unstable or uncompensated respiratory,cardiac,liver,renal diseases.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-07 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 6 months
  A duration from randomization date to disease progression(as defined by RECIST) or death. If a participant
  are known to have progressed, the time to progression is defined as the time from the date of randomization to the date of progression. Otherwise, a participant will be censored at the last date they are known not to be progressed.

SECONDARY OUTCOMES:
Overall survival | 12 months
  Overall Survival is assessed via calculation of the time to death due to any cause. If a participant is known to have died, the time to death is defined as the time from the date of randomization to the date of death. Otherwise, a participant will be censored at the last date they are known to be alive.

CONTACTS AND LOCATIONS:
Overall Officials: Zhang Yi Ping, M.D., Principal Investigator — Zhejiang Cancer Hospital
Locations (6):
- China (6):
  - Hunan Province Tumor Hospital, Changsha, Hunan
  - Sir Run Run Shaw Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Medical School of Zhejiang University, Hangzhou, Zhejiang
  - The Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang